CLINICAL TRIAL: NCT02752100
Title: Long-term Prognosis of Interventional Therapy in Patients With Lower Extremity Arterial Occlusive Disease and Its Risk Factors
Brief Title: A Study on the Effects of Interventional Therapy in Patients With Lower Extremity Arterial Occlusive Disease and Its Risk Factors(EILRF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, MD, PhD, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EILRF
Record Dates: First submitted 2016-03-17; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: PAD
Keywords: Lower Extremity Arterial Occlusive Disease; Interventional Therapy
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional Therapy (Experimental): Percutaneous transluminal angioplasty.
  Interventions: Procedure: Percutaneous transluminal angioplasty
- Non-Interventional Therapy (No Intervention)

INTERVENTIONS:
Procedure: Percutaneous transluminal angioplasty
  Arms: Interventional Therapy

SUMMARY:
Along with the improvement of living standard, the prevalence of Lower extremity arterial occlusive disease (LEAOD) is also increasing, which has become an important cause of lower extremity amputation and greatly affected the patients' life quality. Currently, percutaneous transluminal angioplasty (PTA), including balloon dilatation and stent implantation, has been regarded as the most widely applied and accepted treatment for LEAOD. The therapeutic effects of lower extremity interventional treatment, varied in different reports. It was reported that the therapeutic effects were influenced by some traditional risk factors, including age, gender, smoking, and so on. More risk factors are still unknown. The difference of therapeutic effects, the endpoint events were compared between interventional and conventional treatment group to analyze the effect of interventional treatment on LEAOD and explore its risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 40-90 years old.
* Ankle-brachial index(ABI)<0.9.
* Lower extremity arterial CT shows that the arterial stenosis>50%

Exclusion Criteria:

* Type 2 diabetes with acute complications.
* Type 1 diabetes.
* Cerebrovascular diseases in the last 3 months.
* Cardiovascular diseases (myocardial infarction, angina, cardiac failure) in the last 3 months.
* Hemorrhagic disease.
* Hypohepatia (AST or AST is twice higher than the upper limit) or cirrhosis, hepatic encephalopathy.
* History of dialysis.
* Chronic obstructive pulmonary disease (COPD), chronic respiratory failure or hypoxemia.
* Acute infections, tumor, severe arrhythmia, mental disorders, alcohol or medicine addiction.
* Fertile woman without contraceptives.
* Allergic to iodine.
* Unable to understanding and follow the study protocol orientations.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Ankle-brachial index | Change from baseline at 1 year(End of Trial)
Mortality(%) | 1 year(End of Trial)
Incidence of amputation(%) | 1 year(End of Trial)

SECONDARY OUTCOMES:
Incidence of major adverse cardiac events (MACE)(%) | 1 year(End of Trial)
High-sensitive C reactive protein(mg/L) | Change from baseline at 1 year(End of Trial)
Fasting plasma glucose(mmol/L) | Change from baseline at 1 year(End of Trial)
Blood pressure(mmHg) | Change from baseline at 1 year(End of Trial)
HbA1c(%) | Change from baseline at 1 year(End of Trial)
triglyceride(mmol/L) | Change from baseline at 1 year(End of Trial)
total cholesterol(mmol/L) | Change from baseline at 1 year(End of Trial)
LDL-c(mmol/L) | Change from baseline at 1 year(End of Trial)
HDL-c(mmol/L) | Change from baseline at 1 year(End of Trial)
The lower limb transcutaneous oxygen pressure(mmHg) | Change from baseline at 1 year(End of Trial)

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Liu X, Li Q, Liu Y, He H, Wang K, Yan Z. Quantitative model for assessment of lower-extremity perfusion in patients with diabetes. Med Phys. 2023 May;50(5):3019-3026. doi: 10.1002/mp.16214. Epub 2023 Jan 16. PMID 36617729